CLINICAL TRIAL: NCT06434831
Title: Evaluation of Autonomic Nervous System Changes in Response to Stimulation by Sacral Neuromodulation
Acronym: ESTIME
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023_195
Record Dates: First submitted 2024-03-22; First posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-03

CONDITIONS: Bladder Hyperactivity; Sacral Neuromodulation
Keywords: Bladder hyperactivity; autonomic nervous system; sacral neuromodulation; urodynamic assessment; heart rate variability
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Equipment and Supplies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ANI will be recorded during the SNM. (Experimental)
  Interventions: Device: Medical device for SNM: Interstim II, Interstim micro

INTERVENTIONS:
Device: Medical device for SNM: Interstim II, Interstim micro — ANI will be used during the SNM (2 hours)

SUMMARY:
Overactive bladder syndrome (OAB) is defined by urgent and frequent urges to urinate associated with frequent night-time urination and sometimes urinary incontinence. Sacral neuromodulation (SNM) is now one of the second-line treatments for OAB.

The mode of action of SNM is still poorly understood but a number of data from recent scientific literature suggest that SNM may act, among other things, by altering the balance of the autonomic nervous system (ANS) - located at the interface between the urinary tract and the brain structures regulating the functioning of the urinary tract.

The aim of this study would therefore be to develop a predictive tool for the effectiveness of SNM.

ELIGIBILITY:
Inclusion Criteria:

* Male of female ≥ 18 years
* OAB syndrome
* Indication for a two-staged SNM
* Under general anaesthesia with Remifentanil and Propofol
* Patient who has given written consent to participate in the trial
* Patient willing to comply with all study procedures and duration

Exclusion Criteria:

* Tibial neuro-stimulation (last 3 months)
* Sacral neuromodulation (last 3 months)
* Botulinum toxin A intra-detrusor injection (last 9 months)
* Pregnancy in progress
* Administrative reasons
* Guardianship/curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-07-02 (Estimated); Primary Completion 2026-12-02 (Estimated); Study Completion 2026-12-02 (Estimated)

PRIMARY OUTCOMES:
Comparison of HFVI analysed through HRV at baseline and during standardized stimulation protocol randomly delivered at the level of the 4contact points of the quadripolar lead at the time of lead implantation between the effective and noneffective groups | 1 year
  Comparison of HFVI (high frequence variability index) analysed through heart rate variability (HRV) at baseline and during a standardized stimulation protocol (14 Hz, 210 mcs, amplitude to elicit anal motor response) randomly delivered at the level of the 4 contact points of the quadripolar lead at the time of lead implantation, between the effective and non-effective groups.

SECONDARY OUTCOMES:
Comparison of other HRV parameters at baseline and during a standardized stimulation protocol randomly delivered at the level of the 4 contact points of the quadripolar lead at the time of lead implantation | 1 year
  Comparison of other HRV parameters (SDNN, RMSSD, HF, LF) at baseline and during a standardized stimulation protocol (14 Hz, 210 mcs, amplitude to elicit anal motor response) randomly delivered at the level of the 4 contact points of the quadripolar lead at the time of lead implantation,

IPD SHARING:
Plan to Share IPD: No